CLINICAL TRIAL: NCT01183767
Title: Sunphenon Epigallocatechin-Gallate (EGCg) in Duchenne Muscular Dystrophy
Acronym: SUNIMUD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Friedemann Paul, PI, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUNIMUD
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Epigallocatechin-Gallate; Green tea extract
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGCG (Active Comparator): Epigallocatechin-Gallate (EGCG)
  Interventions: Drug: Epigallocatechin-Gallate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epigallocatechin-Gallate — EGCG in a dosage of up to 10mg/kg body weight
  Arms: EGCG
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this multicentre, prospective, double blind, placebo controlled, randomized pilot study is to investigate safety and tolerance of Epigallocatechin-Gallate (EGCG, the major polyphenol in green tea) in patients with muscular dystrophy of the Duchenne type.

In a second step the investigators want to investigate the effect of EGCG on the course of the Duchenne condition.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is the most frequent neuromuscular condition to occur in childhood and youth. The course of the disease is progressive, and life expectancy is severely curtailed by the participation of the respiratory muscles and/or by progressive cardiomyopathy.

DMD derives from mutations in the DMD gene which leads to a loss of the protein dystrophin. Secondary inflammatory/immunological reactions contribute to the progressive course of the disease (1,2).

No curative therapy yet exists. Administration of steroids is the only established medical treatment. Symptomatic measures are also available, such as orthopaedic operations, the treatment of cardiomyopathy or, in advanced stages, home mechanical ventilation.

In studies involving experiments on cells and animals, Epigallocatechin-Gallate (EGCG, the major polyphenol in green tea) has shown a neuroprotective effect. The neuroprotective mechanism of action is probably based on several factors, including EGCG's modulation of several signal transduction pathways, its influence on the expression of genes regulating cell survival or programmed cell death, as well as its modulation of mitochondrial function.

The mdx mouse is the best-investigated animal model of a dystrophin-negative muscular dystrophy. Administration of EGCG in the mdx mouse led to both a reduction in the proportion of fibre necroses as well as to a less pronounced proliferation of connective tissue in the muscle (3,4), and also to an improvement in clinical symptoms (5,6).

Therefore, the investigators want to investigate safety and tolerance of EGCG in a dosage of up to 10mg/kg in patients with muscular dystrophy of the Duchenne type in this multicentre, prospective, double blind, placebo controlled, randomized pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy
* age 5-10 years
* ability to walk without support
* informed consent by the parents

Exclusion Criteria:

* another serious organic disease
* further primary psychiatric or neurological diseases
* long-term intake of liver-toxic medicines

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2010-12-30 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 12 months
  safety and tolerability in terms of number of adverse events in which a causal relationship with the test substance cannot be excluded, and GLDH values.

SECONDARY OUTCOMES:
efficacy | 36 months
  changes in the means of the 6 minute walk test (baseline to visit after month 36).

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Dr., Study Director — Charite University, Berlin, Germany
Locations (3):
- Germany (3):
  - Charité University Berlin, Berlin
  - DRK Kliniken Berlin, Westend, Pädiatrie, Berlin
  - Diakonisches Werk Oldenburg SPZ, Oldenburg